CLINICAL TRIAL: NCT04322006
Title: A Phase I/II Study of Evaluating the Safety, Tolerance, Pharmacokinetics, Pharmacodynamics and Curative Effect of Dose Escalation and Extension for Single Drug TJ004309 and Toripalimab Combine Treatment for Advanced Solid Tumor
Brief Title: A Phase I/II Study of TJ004309 for Advanced Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ004309STM102
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ004309 injection Monotherapy or Combination with Toripalimab (Experimental): TJ004309 will be dose escalated in a 3+3 design in Monotherapy or combination with Toripalimab
  Interventions: Drug: TJ004309; Drug: Toripalimab

INTERVENTIONS:
Drug: TJ004309 — Antibody to CD73
Drug: Toripalimab — Humanized monoclonal antibody to PD-1

SUMMARY:
This study is a phase I/II study of single drug TJ004309 and Toripalimab combine treatment for Advanced solid tumor. This study include two stages. First stage is dose escalation and second stage is dose extension. The purpose of part A is to confirm the MTD or MED and the clinical dose. The purpose of part B is to observe the safety, effectiveness, Pharmacokinetics, pharmacodynamics and biomarker properties for effective subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* In the dose-escalation phase, subjects with advanced solid tumors that are histologically or cytologically confirmed to be unresectable or have metastasized, subjects with standard treatment failure or intolerance (disease progression, or inability to tolerate chemotherapy, targeted therapy, etc.), or subjects without effective treatment.
* Synchronous dose expansion (will base on dose-escalation phase)
* At least one measurable disease by modified RECIST 1.1 for immune based therapeutics V1.1
* Expected survival ≥ 3 months
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 times upper limit of normal (ULN)
  * Total serum bilirubin ≤ 1.5 times the ULN
  * Absolute neutrophil count (ANC) ≥ 1.5 ×109/ L
  * Platelets ≥ 100×109/ L without transfusion support within 28 days prior to study treatment
  * Hemoglobin ≥ 9.0 g/dL without transfusion support within 14 days prior to study treatment
  * Serum creatinine ≤ 1.5 times the ULN or Creatinine clearance > 30 mL/min by Cockcroft-Gault formula
  * International normalized ratio (INR) in normal range
* Serum pregnancy test must be negative for childbearing female prior to study treatment
* The man have reproductive ability or childbearing female (refers to men and women not on birth control operation, and the menopause women), must use the highly effective contraceptive methods (such as oral contraceptives, intrauterine contraceptive device, abstemious sexual desire or barrier contraceptive method combined with spermicide) during the study, and sustain contraception 6 months after the last dose
* Willingness and ability to consent for self to participate in study and comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Pregnancy or breastfeeding
* Prior T-cell therapy
* Receipt of systemic anticancer therapy or ≥ 5 times the elimination half-life of the drug has elapsed within 2 weeks prior to study treatment (Note: whichever is shorter shall prevail.)
* Exist ≥ 2 kinds of primary tumor, expect cured preinvasive carcinoma and basaloma. (patients are not excluded if ≥ 5 years treatment with other tumor prior to study treatment.)
* Autoimmune disease requiring treatment within the past twelve months only requiring related treatment replacement
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications more than 7 days within 14 days prior to study treatment (Note: inhaled and topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.)
* Current treatment on another therapeutic clinical trial within 14 days prior to study treatment
* Major surgical procedure or significant traumatic injury within 4 weeks prior to study treatment and no date of surgery (if applicable) or anticipated need for a major surgical procedure planned during study treatment
* Chest radiotherapy ≤ 4 weeks, wide field radiotherapy ≤ 4 weeks (defined as > 50% of volume of pelvic bones or equivalent) or palliative radiotherapy ≤ 2 weeks prior to study treatment
* Brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease, unless the lesion(s) have been radiated or resected, are considered fully treated and inactive, are asymptomatic, and no steroids have been administered for central nervous system disease over the 2 weeks prior to study treatment
* Known active viral or nonviral hepatitis or cirrhosis, except patients with Hepatitis C infection and undetectable virus following treatment are eligible.
* Known human immunodeficiency virus (HIV) positive
* Ascites or pericardial effusion that can not be control
* History of or active interstitial lung disease
* Hypertension is not well controlled by medication. Hypertension defined as blood pressure (BP) systolic > 150 or diastolic > 90 mm Hg (Note: Initiation or adjustment of antihypertensive medication prior to study entry is allowed provided that the average of the three most recent BP readings prior to study enrollment is ≤150/90 mm Hg.)
* Cardiovascular diseases with clinical significance, include phase II-III cardiac insufficiency defined by New York Heart Association, myocardial infarction (MI) within 3 months prior to study treatment, symptomatic congestive heart failure, cerebral infarction within 3 months prior to study treatment, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) within 6 months prior to study treatment
* Deep-venous thrombosis within 6 months prior to study treatment (except treated without warfarin 2 weeks prior to study treatment)
* Thrombolytic use (except to maintain IV catheters) within 10 days prior study treatment
* Any active infection requiring systemic treatment
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities(DLT) | 28days after first dose for QW, 21days after first dose for Q3W
  The safety and tolerance of TJ004309
MTD | 2 years
  Maximum tolerated dose (MTD)
MED | 2 years
  Maximum effective dose (MED)
Recommend dose of TJ004309 | 2 years
  Recommend dose of TJ004309

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Cancer Hospital affiliated to Shantou University Medical College, Shantou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang